CLINICAL TRIAL: NCT07133490
Title: Intraperitoneal Irinotecan Combined With Systemic Therapy for Patients With Gastric Peritoneal Metastases: A Phase II, Multicenter Study
Brief Title: INTERACT Stomach-II
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); Netherlands Cancer Institute - NKI (Unknown)
Responsible Party: Principal Investigator, Pieter Christiaan van der Sluis, Dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-521468-36-00; 2025-521468-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-06; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Peritoneal Metastases From Gastric Cancer
Keywords: Gastric cancer; Peritoneal metastases; Intraperitoneal chemotherapy; Irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraperitoneal chemotherapy arm (Experimental): Patients in this group will receive intraperitoneal irinotecan in addition to standard systemic therapy
  Interventions: Drug: intraperitoneal chemotherapy

INTERVENTIONS:
Drug: intraperitoneal chemotherapy — Through a peritoneal access port, irinotecan will be administered at the same time as systemic (chemo)therapy

SUMMARY:
This is a phase II study conducted in three hospitals in the Netherlands (Erasmus MC in Rotterdam, Catharina Hospital in Eindhoven, and the Netherlands Cancer Institute in Amsterdam). A total of 49 patients will take part. The aim is to test whether a new combination treatment is feasible for patients with gastric peritoneal metastases (PM). The treatment includes chemotherapy (intraperitoneal irinotecan and standard systemic therapy such as CAPOX or FOLFOX), and may also include nivolumab or trastuzumab, depending on biomarker results.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer or gastroesophageal junction adenocarcinoma
* Pathologically and clinically confirmed diagnosis of macroscopic peritoneal metastases (defined as PCI score ≥ 1)
* WHO-performance score of 0 to 1 with a life expectancy greater than or equal to three months
* Aged 18 years or older
* Written informed consent according to the ICH-GCP and national/local regulations

Exclusion Criteria:

* Distant metastases other than peritoneal metastases or metastatic lymph nodes
* Prior palliative systemic therapy for gastric cancer
* Prior (neo)-adjuvant systemic therapy for gastric cancer within the six months before enrolment in this study
* Severe symptomatic ascites requiring monthly recurrent therapeutic paracentesis
* Homozygous dihydropyrimidine dehydrogenase (DPD) deficiency
* Any contra-indication for the (planned) systemic chemotherapy (e.g. active infection, serious concomitant disease, severe allergy, persistent neurologic toxicity after (neo-)adjuvant oxaliplatin based systemic therapy), as determined by the treating medical oncologist
* Inadequate organ functions (defined as a hemoglobin <5.0 mmol/l, an absolute neutrophil count <1.5 x 109/l, platelet count <100 x 109/l, creatinine clearance <30 ml/min, bilirubin >2x ULN and liver transaminases >2.5x ULN)
* Pregnant or lactating women
* Concomitant participation in any clinical study that could modify the outcomes relevant to this study
* Absence of assurance of compliance with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intraperitoneal administration of irinotecan | From enrollment until the completion of all chemotherapy cycles: either 6 cycles of CAPOX (21 days per cycle) or 8 cycles of FOLFOX (14 days per cycle)
  Percentage of patients who completed all planned cycles of intraperitoneal irinotecan in combination with systemic therapy (6 cycles in the case of CAPOX, 8 cycles in the case of FOLFOX)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter C van der Sluis, MD PhD, Principal Investigator — Erasmus MC, University Medical Center Rotterdam

IPD SHARING:
Plan to Share IPD: No